CLINICAL TRIAL: NCT01712958
Title: Quantifying Micro RNA Levels to Obtain a Micro RNA Signature of Colon Tumor Phenotypes and Sub Phenotypes
Brief Title: Quantifying Micro RNA Levels of Colon
Acronym: CRC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0148
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Carcinoma (CRC) Patients
Keywords: CRC miRNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: human colon and rectal tumors, tumor adjacent and normal tissues
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer and the fourth leading cause of cancer-related death in the world. Despite potentially curative surgery and the use of modern adjuvant chemotherapy, up to 40% of CRC patients subsequently develop local tumor relapse or metastatic disease. Currently, aside from post-operative pathological staging, early follow up of the patients does not include a specific test or any other evaluation that could predict disease recurrence. Therefore, exploring and identifying novel biomarkers of CRC's following diagnosis of the primary tumor may help us in identifying patients at high risk for recurrence.

Modifications in signaling pathways and their regulation by microRNAs (miRNAs) are being evaluated as biomarkers and therapeutic targets for cancer in general and CRC in particular. It has been established, although not completely, that miRNAs have a role in initiation and progression of CRC. Modifications of miRNAs have been recorded in CRC tumors, and the expression patterns of these miRNAs could in principle biomark this cancer's phenotype. As miRNAs are well documented to regulate critical molecules in signaling pathways, their regulation of tumor relevant pathways may also serve to further sub-classify patients into drug responsive groups. Moreover, miRNAs may be sampled from peripheral blood and are available as a non-invasive diagnostic method, their application as biomarkers is of special interest.

In this study the investigators aim to quantify miRNA levels in human colon and rectal tumors, tumor adjacent and normal tissues. By comparing this data from a large cohort of patients, the investigators aim to identify specific, relevant miRNAs that may serve as biomarkers to stratify CRC patients according to their clinical characteristics such as disease stage, specific treatment, prognosis and disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

Adult men and women over the age of 18 years who underwent colon resection of any kind are suitable candidates for this study.

Exclusion Criteria:

Pregnant woman and children (under the age of 18 years) will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CRC patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
identifying specific, relevant miRNAs that may serve as biomarkers to stratify CRC patients according to their clinical characteristics | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Avital, M.D., Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel